CLINICAL TRIAL: NCT06969339
Title: Unilateral Posterior Wedge Closing Vertebral Column Resection for Treatment of Adolescent Neglected Congenital Kyphoscoliosis
Brief Title: Unilateral Posterior Wedge Closing Vertebral Column Resection for Treatment of Congenital Kyphoscoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Eissa Moussa, resident at the Orthopaedic and Trauma Surgery department, Assiut University
Other Study IDs: Posterior wedge closing
Record Dates: First submitted 2025-05-02; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Unilateral Posterior Wedge Closing
Keywords: unilateral posterior wedge closing; neglected congenital kyphoscoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with untreated congenital kyphoscoliosis, no prior surgery: adolescent patients with untreated congenital kyphoscoliosis, no prior surgery, and complete imaging/follow-up data.

SUMMARY:
A retrospective analysis of 12 adolescents undergoing unilateral posterior wedge closing VCR for neglected congenital kyphoscoliosis, assessing surgical outcomes over a mean 2.9-year follow-up.

DETAILED DESCRIPTION:
Design: Single-center case series (Assiut University Hospital, 2015-2020).

Intervention: Modified posterior VCR with unilateral convex wedge resection, spinal shortening, and instrumentation.

Key Steps:

Preoperative CT/MRI for anatomical planning.

Posterior-only approach with pedicle screw instrumentation.

Wedge resection focused on convex side, preserving concave continuity.

Bone grafting (cancellous or mesh cage) post-correction.

Follow-up: Radiographic and clinical assessments up to 2 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

Age >10 years.

Congenital kyphoscoliosis diagnosis.

No prior spinal surgery.

Preoperative CT/MRI and 24-month follow-up data.

Exclusion Criteria:

Idiopathic or neuromuscular scoliosis

Previous spinal surgery

Incomplete radiographic or follow-up data

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consisted of adolescents (mean age 15.7 years) with neglected congenital kyphoscoliosis, who had not undergone any prior spinal surgery and had complete preoperative and follow-up imaging data. The sample represents a total coverage of all cases meeting criteria during the study period, reflecting the rarity of congenital kyphoscoliosis requiring surgical intervention in adolescence, The patients who have moderate to severe spinal deformity, with a mean preoperative Cobb angle of 53.2° (kyphoscoliosis involves abnormal curvature in both sagittal and coronal planes, hese cases typically present during adolescence, coinciding with the second growth spurt, which is a known period for progression of congenital spinal deformities
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cobb angle correction | Baseline, and 2-year follow-up.
  Change in coronal deformity angle (pre-op to post-op and 2-year follow-up).

SECONDARY OUTCOMES:
Blood loss | Intraoperative
  Intraoperative hemorrhage volume.

REFERENCES:
- [Background] Suk SI, Kim JH, Kim WJ, Lee SM, Chung ER, Nah KH. Posterior vertebral column resection for severe spinal deformities. Spine (Phila Pa 1976). 2002 Nov 1;27(21):2374-82. doi: 10.1097/00007632-200211010-00012. PMID 12438987
- [Background] Yang JH, Kim HJ, Chang DG, Suh SW, Nam Y, Hong JY. The Efficacy of Single-Stage Correction by Posterior Approach for Neglected Congenital Scoliosis: Comparative Analysis According to the Age of Surgical Intervention. J Clin Med. 2022 Apr 19;11(9):2278. doi: 10.3390/jcm11092278. PMID 35566404